CLINICAL TRIAL: NCT02346708
Title: Cortical Physiology as a Therapeutic Target in Parkinson's Disease Related Dementia and Cognitive Dysfunction
Brief Title: Cognitive Dysfunction in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-2724; 1K02NS080885-01A1 (NIH)
Record Dates: First submitted 2015-01-09; First posted 2015-01-27 (Estimated); Results first posted 2020-12-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's; TMS; Kluger
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real TMS (Experimental): TMS will be administered using a 70-mm diameter air-cooled figure-of-8 coil and SuperRapid2 Magstim Stimulator. Repetitive pulses will be delivered to the right and left pre-frontal cortex (Brodmann area 46) using a frameless stereotactic navigation system and the subject's magnetic resonance imaging (MRI) in Brainsight software. Stimuli will be delivered at 20 Hz at 90% resting motor threshold (rMT) for 25 trains of 30 pulses per train, inter-train interval of 30 seconds for a total of 750 pulses per hemisphere. This dose and duration of repetitive TMS (rTMS) is based on physiological studies of healthy adults and treatment studies of cognition in PD and Alzheimer's disease.52, 123 Side of first stimulation (left vs right hemisphere) will be counterbalanced across subjects.
  Interventions: Device: Real TMS
- Sham TMS (Sham Comparator): Sham stimulation will be delivered using a sham coil fitted with electrodes to mimic both the auditory and somatic sensation of real TMS.
  Interventions: Device: Sham TMS

INTERVENTIONS:
Device: Real TMS — real treatment
  Other Names: Transcranial Magnetic Stimulation
  Arms: Real TMS
Device: Sham TMS — placebo treatment
  Arms: Sham TMS

SUMMARY:
This study plans to learn more about the brain function related to thinking problems in individuals with Parkinson's disease.

DETAILED DESCRIPTION:
Dementia is the leading cause of nursing home placement in Parkinson's disease (PD) yet little is known about the cause(s) of cognitive dysfunction in PD and there are no effective treatments. The investigators preliminary data and other published studies suggest that abnormalities in brain activity involving networks important for normal thinking and memory may contribute to cognitive dysfunction in PD and may represent a target for treatment. This proposal will identify abnormalities in cortical activity related to cognitive dysfunction in PD using magnetoencephalography and will perform a randomized control trial of bifrontal repetitive transcranial magnetic stimulation to determine the therapeutic potential of modulating this brain activity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable PD (using United Kingdom Brain Bank criteria)
* Diagnosis of mild cognitive impairment
* No unstable medical condition

Exclusion Criteria:

* Features suggestive of other causes of Parkinsonism or other neurological disorders
* Prior deep brain stimulation (DBS) or ablation surgery
* Evidence for active depression or Hospital Anxiety and Depression Scale (HADS) score greater than or equal to 11
* Motor symptoms expected to interfere with scanning (e.g. sever tremor)
* Contraindications to TMS, MEG, or MRI such as pregnancy, pacemaker, unstable cardiac disease, skull lesion, claustrophobia, history of epilepsy, or on medications known to lower seizure threshold
* Implanted electronic devices or metal

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-01; Primary Completion 2018-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benzi M Kluger, MD, MS, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado School of Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available to the scientific community upon request.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted in the United States at one site: University of Colorado Denver - Anschutz Medical Campus. The first participant was enrolled in May 19, 2014.
Pre-assignment Details: 70 participants were assessed for eligibility (following Inclusion and exclusion criteria), 21 were screen failures, 49 participants were randomized to treatment.
Groups:
- Real TMS: TMS will be administered using a 70-mm diameter air-cooled figure-of-8 coil and SuperRapid2 Magstim Stimulator. Repetitive pulses will be delivered to the right and left dorsolateral pre-frontal cortex (Brodmann area 46) using a frameless stereotactic navigation system and the subject's magnetic resonance imaging (MRI) in Brainsight software. Stimuli will be delivered at 20 Hz at 90% resting motor threshold (rMT) for 25 trains of 30 pulses per train, inter-train interval of 30 seconds for a total of 750 pulses per hemisphere. This dose and duration of repetitive TMS (rTMS) is based on physiological studies of healthy adults and treatment studies of cognition in PD and Alzheimer's disease. Side of first stimulation (left vs right hemisphere) will be counterbalanced across subjects.
  Real TMS: real treatment
Period: Overall Study
Arm/Group | Real TMS | Sham TMS
Started | 24 | 25
Completed | 22 | 24
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Real TMS: TMS will be administered using a 70-mm diameter air-cooled figure-of-8 coil and SuperRapid2 Magstim Stimulator. Repetitive pulses will be delivered to the right and left dorsolateral pre-frontal cortex (Brodmann area 46) using a frameless stereotactic navigation system and the subject's magnetic resonance imaging (MRI) in Brainsight software. Stimuli will be delivered at 20 Hz at 90% resting motor threshold (rMT) for 25 trains of 30 pulses per train, inter-train interval of 30 seconds for a total of 750 pulses per hemisphere. Stimulation will be delivered for 10 consecutive days, excluding the weekends. This dose and duration of repetitive TMS (rTMS) is based on physiological studies of healthy adults and treatment studies of cognition in PD and Alzheimer's disease. Side of first stimulation (left vs right hemisphere) will be counterbalanced across subjects.
  Real TMS: real treatment
- Total: Total of all reporting groups
Arm/Group | Real TMS | Sham TMS | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 14 | 17 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (7.2) | 69.5 (8) | 68.5 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 16 | 17 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 20 | 24 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change in Magnetoencephalography (MEG) Connectivity Measures
Description: Our MEG outcome will be a change in small-worldness, global efficiency, nodal efficiency and degree distribution pre-TMS to immediately post-TMS treatment.
Time Frame: 2 weeks
Population: No data displayed because Outcome Measure has zero total analyzed. No participants were analyzed for this outcome measure.
Groups:
- Real TMS: TMS will be administered using a 70-mm diameter air-cooled figure-of-8 coil and SuperRapid2 Magstim Stimulator. Repetitive pulses will be delivered to the right and left dorsolateral pre-frontal cortex (Brodmann area 46) using a frameless stereotactic navigation system and the subject's magnetic resonance imaging (MRI) in Brainsight software. Stimuli will be delivered at 20 Hz at 90% resting motor threshold (rMT) for 25 trains of 30 pulses per train, inter-train interval of 30 seconds for a total of 750 pulses per hemisphere. This dose and duration of repetitive TMS (rTMS) is based on physiological studies of healthy adults and treatment studies of cognition in PD and Alzheimer's disease.52, 123 Side of first stimulation (left vs right hemisphere) will be counterbalanced across subjects.
  Real TMS: real treatment
Arm/Group | Real TMS | Sham TMS
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Post-TMS Change From Baseline in Cognitive Scores
Description: Our behavioral outcome will be a change in the scores of the following tests:
  Mattis Dementia Rating Scale: Higher raw scores = better cognitive status, ranging from 0 to 144. Normative data in healthy subjects range from 137 to 144.
  Trail Making Test Trails B: average score is 75 seconds; deficient score is > 273 seconds.
  Delis-Kaplan Executive Function System (DKEFS) - Verbal Fluency Test. Higher score = higher ability in language processing. Scales scores vary from 0 min to N/A max (no concrete maximum).
  DKEFS - Stroop Interference Test measures inhibitory control and cognitive flexibility. Performance is measured by completion time. No min or max value for this test. Test should be discontinued after 90 sec.
  For those, higher scores = higher abilities: California Verbal Learning Test (declarative memory, scale 0 to 80), Boston Naming Test (language, scale 0 to 60), Brief Test of Attention and Judgment of Line Orientation (scale 0 to 30)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Real TMS | Sham TMS
Number analyzed (Participants) | 22 | 24
Scores on a scale
  Score on the Mattis Dementia Rating Scale (MDRS) at 2 weeks minus score on the MDRS at baseline | -1.4 (4.55) | 0 (5.55)
  Score on the Verbal fluency at 2 weeks minus score on the Verbal fluency at baseline | 0.3 (11.35) | 1 (15.7)
  Score on the Stroop Interference at 2 weeks minus score on the Stroop Interference at baseline | -9.1 (18.55) | -2.9 (18.85)
  Score on the Brief Test of Attention (BTA) at 2 weeks minus score on the BTA at baseline | -0.1 (4) | 0.6 (4.15)
  Score on the Boston Naming Test (BNT) at 2 weeks minus score on the BNT at baseline | 0.2 (5.95) | 1.4 (2.25)
  Score on the Judgment of Line Orientation (JLO) at 2 weeks minus score on the JLO at baseline | 0.9 (4.7) | 1 (4.2)
Statistical Analysis 1: Comparison: Real TMS vs Sham TMS; We estimated a sample size of 20 per group would provide at least 80% power at a significance level of 0.05 to detect a between-group difference of 10 on the Matthis Dementia Rating Scale-2, an effect size similar to prior studies of rivastigmine; Test type: Superiority; p = 0.1, Mixed Models Analysis — We determined whether there was a significant group difference between the real and sham treated PD-MCI patients on the DRS-2 change following rTMS using mixed model regression (MMR) to fit longitudinal models; degrees of freedom: 46; Mean Difference (Final Values) = -2.07, 95% CI 2-sided [-4.56 to 0.42]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the study, i.e. 6 weeks.
Groups:
- Real TMS: TMS will be administered using a 70-mm diameter air-cooled figure-of-8 coil and SuperRapid2 Magstim Stimulator. Repetitive pulses will be delivered to the right and dorsolateral left pre-frontal cortex (Brodmann area 46) using a frameless stereotactic navigation system and the subject's magnetic resonance imaging (MRI) in Brainsight software. Stimuli will be delivered at 20 Hz at 90% resting motor threshold (rMT) for 25 trains of 30 pulses per train, inter-train interval of 30 seconds for a total of 750 pulses per hemisphere. This dose and duration of repetitive TMS (rTMS) is based on physiological studies of healthy adults and treatment studies of cognition in PD and Alzheimer's disease. Side of first stimulation (left vs right hemisphere) will be counterbalanced across subjects.
  Real TMS: real treatment
Arm/Group | Real TMS | Sham TMS
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/24
Other Adverse Events (participants affected / at risk) | 6/22 | 1/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real TMS (N=22) | Sham TMS (N=24)
Hospitalization (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real TMS (N=22) | Sham TMS (N=24)
vasovagal syncope (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
local pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
motor problems (Nervous system disorders) | 0 (0) | 1 (1)
mild blurry vision (Eye disorders) | 1 (1) | 0 (0)
confusion (Nervous system disorders) | 0 (0) | 1 (1)
burst vein in eye (Vascular disorders) | 1 (1) | 0 (0)
mild flu (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Our specialized MEG data analyst working on the Primary outcome has encountered a Covid-related family emergency, which has delayed the analysis process.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-23): https://cdn.clinicaltrials.gov/large-docs/08/NCT02346708/Prot_SAP_000.pdf